CLINICAL TRIAL: NCT04263597
Title: Oral Supplementation of 2'-Fucosyllactose in Allogeneic Bone Marrow Transplant Recipients to Maintain Intestinal Homeostasis
Brief Title: Oral Supplementation of 2'-Fucosyllactose in Allogeneic Bone Marrow Transplant Recipients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-0008
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic Stem Cell Transplant
MeSH Terms: interventions — 2'-fucosyllactose

STUDY DESIGN:
Intervention Model Description: Eligible patients will be allocated into the following arms as determined by age at enrollment.
  Arm 1: 0-5 years; Arm 2: 5.1-10 years; Arm 3: >10 years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 2'-fucosyllactose for ages 0-5 years (Experimental): Dose for ages 0-5 years: 2.5 g/day;
  Interventions: Drug: 2'-fucosyllactose
- 2'-fucosyllactose for ages 5.1-10 years (Experimental): Dose for ages 5.1-10 years: 5 g/day;
  Interventions: Drug: 2'-fucosyllactose
- 2'-fucosyllactose for ages >10 years (Experimental): Dose for ages >10 years: 10 g/day;
  Interventions: Drug: 2'-fucosyllactose

INTERVENTIONS:
Drug: 2'-fucosyllactose — 2FL powder will be provided to participants randomized to receive 2FL in packets. They will be instructed to drink this daily by adding the required amount to food or drink. It may also be mixed in standard feeds or mixed with water and administered by enteral tube, whenever applicable.
  Other Names: 2FL supplementation

SUMMARY:
High dose chemotherapy and radiation used as preparative regimens in patients undergoing an allogeneic hematopoietic stem cell transplant (HSCT) disrupts intestinal homeostasis by damaging the intestinal epithelium and altering the intestinal microbiome. The investigators hypothesize that 2'-fucosyllactose (2FL) supplementation will be safe and tolerable and result in an increase in the relative abundance of intestinal Bifidobacteria. The investigators also hypothesize that 2FL supplementation will lead to reduction of Firmicutes and/or Proteobacteria, and improved intestinal homeostasis at day+30 as measured by lower pro-inflammatory cytokines, reduced levels of T-cell activation, lower markers of intestinal injury (fecal human DNA and plasma reg-3-alpha), increased fecal butyrate levels and ultimately lower incidence of acute GVHD and BSI at day+100.

Phase II:

The investigators hypothesize that 2FL supplementation will be safe and tolerable and result in an increase in the relative abundance of fecal short chain fatty acids such as butyrate, acetate and propionate at day+7 compared to baseline values.

DETAILED DESCRIPTION:
This phase I/IIa study is a single center prospective study at Cincinnati Children's Hospital Medical Center (CCHMC).

This study will assess the safety and tolerability of various doses of 2FL. Eligible patients will be allocated to the following arms as determined by age at enrollment:

Arm 1: 0-5 years; Arm 2: 5.1-10 years; Arm 3: >10 years

The investigators will first enroll 5 patients of ages ≥10 years undergoing allogeneic HSCT. 2'-FL will be administered to these patients from day-7 until day+30 after HSCT at the starting dose for the ≥10 years age group. Once safety is determined the investigators will then enroll an additional 5 patients of ages 5-10 years and 5 patients of ages 0-5 years and administer 2'FL at starting doses according to their age group to children from day-7 to day+30 after HSCT. Enrollment in the 2 defined age groups (5-10 years and 0-5 years) will occur independent of each other/in parallel to establish safety. Once safety is established in these patients the investigators will proceed with the 3x3 study design dose finding portion of our study

Three patients will be enrolled in each arm at the starting dose level. Investigators will perform a dose escalation or de-escalation based on rates of dose limiting toxicities.

Phase II:

Initial 15 patients to establish safety as per the FDA have been enrolled. An additional 10 patients were enrolled and interim analyses demonstrating safety, lack of any dose limiting toxicities and a positive signal of increase in fecal acetate and propionate at day+7 compared to baseline values) were performed. The investigators will enroll approximately 65 additional patients to test efficacy of 2FL supplementation in children and young adult allogeneic HSCT patients with a goal to reduce intestinal inflammation and improve post HSCT outcomes such as acute GVHD and bloodstream infections.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled for allogeneic stem cell transplant
* All ages and underlying diagnoses, preparative regimens, stem cell sources and acute GVHD prophylaxes

Exclusion Criteria:

* Unable to take anything orally or enterally (i.e. intestinal failure)
* Actively breastfeeding infants
* Recent (within the week prior to enrollment) GI infection
* Patients receiving anti-diarrheal medications such as loperamide
* Patients who have received probiotics or prebiotics during the previous month
* Patients who have had any type of gut damage within the past 3 months such as previous bowel perforations, previous episode of Grade 4 neutropenic colitis or typhlitis
* Patients with inflammatory bowel disease, short bowel syndrome, and patients with a history of bowel resections

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Number of bloodstream infections | Day+100 after transplant
  Number of bloodstream infections in patients on 2FL
Number of patients able to take 2FL | 1 week prior to start of chemotherapy until day+30 after transplant
  6 of 10 patients receiving 2FL able to take 80% of their planned doses
Change in fecal butyrate/acetate/propionate levels | Day+ 7 after transplant
  Change in fecal butyrate/acetate/propionate levels from baseline at day+ 7 in patients enrolled in phase II of the study

SECONDARY OUTCOMES:
Relative abundance of fecal Bifidobacteria at day+30 compared to baseline by >/=10% | Day+30 after transplant
  Change in relative abundance of fecal Bifidobacteria at day+30 compared to baseline by >/=10%
Relative abundance of fecal Firmicutes and Proteobacteria at day+30 compared to baseline for patients on 2FL | Day+30 after transplant
  Change in relative abundance of fecal Firmicutes and Proteobacteria at day+30 compared to baseline for patients on 2FL
Incidence of acute GVHD | Day+100 after transplant
  Incidence of acute GVHD in patients on 2FL
Incidence of bloodstream infections | Day+100 after transplant
  Incidence of bloodstream infections in patients on 2FL
Incidence of mucosal barrier injury laboratory-confirmed bloodstream infection (MBI-LCBI) | Day+ 100 after transplant
  Incidence of MBI-LCBI in patients enrolled in phase II of the study
Incidence of graft versus host disease (GVHD) | Day+ 100 after transplant
  Incidence of GVHD in patients enrolled in phase II of the study
Urine 3-indoxyl sulfate (3-IS) Levels | Baseline, day+7, day+14, day+30 after transplant
  Urine 3-IS levels at day+7/day+14/day+30 compared to baseline in patients enrolled in phase II of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Khandelwal, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No